CLINICAL TRIAL: NCT03333564
Title: Effect of Vitamin D3 and Omega-3FA on Estradiol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science Private University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DRGS-2014-2015-165
Record Dates: First submitted 2017-10-27; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-10

CONDITIONS: Vitamin D Deficiency
Keywords: Vitamin D3; Vitamin D deficiency; estradiol; omega-3 fatty acids; menopausal
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VD3 group (Experimental): treated with 50,000 IU VD3 / week
  Interventions: Dietary Supplement: VD3
- omega3-FA group (Experimental): 1000 mg wild salmon and fish oil complex (contains 300 mg of omega3-FA) once daily
  Interventions: Dietary Supplement: Omega3-FA
- VD3 and Omega-3FA group (Experimental): 50,000 IU VD3 / week and 1000 mg wild salmon and fish oil complex (contains 300 mg of omega-3FA) once daily
  Interventions: Dietary Supplement: VD3 and Omega-3FA
- Control group (Other): No intervention was given
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: VD3 — 50,000 IU VD3 / week for 8 weeks
  Arms: VD3 group
Dietary Supplement: Omega3-FA — 300 mg of omega3-FA once daily for 8 weeks
  Arms: omega3-FA group
Dietary Supplement: VD3 and Omega-3FA — 50,000 IU VD3 / week for 8 weeks and 300 mg of omega-3FA once daily for 8 weeks
  Arms: VD3 and Omega-3FA group
Other: Control — No intervention was given
  Arms: Control group

SUMMARY:
The effect of vitamin D3 and omega-3 Fatty acids on estradiol levels.

DETAILED DESCRIPTION:
The data about effect of vitamin D3 (VD3) and omega-3 fatty acids (omega-3FA) on serum levels of estradiol (E2) are scarce and conflicting and nothing is published in the literature about the effect of the combination of VD3 and omega-3FA on the E2 levels.

This study was conducted to investigate effect of VD3 and omega-3FA alone and with each other on serum E2 levels in premenopausal females with vitamin D deficiency (VDD).

This randomized, placebo-controlled clinical trial was designed to test effects of 50,000 IU VD3 weekly and 300 mg omega-3FA daily for eight weeks, separately and with each other, on the mid-follicular serum levels of E2 and 25-hydroxy vitamin D (25OHD). This study was conducted during winter in 86 healthy premenopausal Jordanian females with VDD with a mean age of (32.8 ± 8.9) years. Fasting serum levels for 25OHD, E2, PTH (parathyroid hormon), calcium, phosphate, ALT (alanine aminotransferase), and urea were assessed at baseline and the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal females
* Medical diagnosis of vitamin D deficiency (VD < 30 ng / ml)

Exclusion Criteria:

* Women previously diagnosed with any chronic disease such as kidney diseases were excluded from the study due to the effect of prolonged administration of VD3 on kidney stones formation. Women who are pregnant, breastfeeding or using hormonal contraceptives were also excluded.

Ages: 22 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Premenopausal females
Enrollment: 116 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Plasma concentrations of 25-hydroxyvitamin D, estradiol | 8 weeks
  Concentration

SECONDARY OUTCOMES:
Plasma concentrations of PTH, Ca | 8 weeks
  Concentration

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud S Abu-Samak, PhD, Principal Investigator — Applied Science Private University

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP
Time Frame: when summary data are published
Access Criteria: open access

REFERENCES:
- [Background] Holick MF, Chen TC. Vitamin D deficiency: a worldwide problem with health consequences. Am J Clin Nutr. 2008 Apr;87(4):1080S-6S. doi: 10.1093/ajcn/87.4.1080S. PMID 18400738
- [Derived] Al-Shaer AH, Abu-Samak MS, Hasoun LZ, Mohammad BA, Basheti IA. Assessing the effect of omega-3 fatty acid combined with vitamin D3 versus vitamin D3 alone on estradiol levels: a randomized, placebo-controlled trial in females with vitamin D deficiency. Clin Pharmacol. 2019 Feb 4;11:25-37. doi: 10.2147/CPAA.S182927. eCollection 2019. PMID 30787641